CLINICAL TRIAL: NCT04528823
Title: GXT - GeneXpert or Chest-X-ray or Tuberculin Skin Testing for Household Contact Assessment: a Cluster Randomized Trial
Brief Title: GXT - GeneXpert or Chest-X-ray or Tuberculin Skin Testing for Household Contact Assessment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Dick Menzies, Senior investigator at Research Institute of Mcgill Unniversity Health Centre, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FND-143350-2
Record Dates: First submitted 2020-07-13; First posted 2020-08-27 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2023-07

CONDITIONS: Latent Tuberculosis
Keywords: Latent Tuberculosis; GeneXpert; Chest X-Ray; Tuberculin Skin Testing
MeSH Terms: conditions — Latent Tuberculosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard care (control arm) (No Intervention): Strategy 1: Symptoms screen, CXR and TST (standard)
- GeneXpert (GX) (Active Comparator): Strategy 2: Symptoms screen, Genexpert and TST
  Interventions: Other: Strategy 2: Symptom screen, Genexpert and TST
- CXR for all/NoTST (Active Comparator): Strategy 3: Symptoms screen, CXR but NO TST
  Interventions: Other: Strategy 3:Symptom screen, CXR but NO TST

INTERVENTIONS:
Other: Strategy 2: Symptom screen, Genexpert and TST — Participants follow an algorithm similar to the standard care, however participants with positive symptom screen and/or positive TST will receive GX (i.e., GX replaces CXR in standard care algorithm). GX positive are considered to have active TB. TST positive and GX negative receive LTBI treatment. If an individual is not able to provide sputum, they will undergo a CXR.
  Arms: GeneXpert (GX)
Other: Strategy 3:Symptom screen, CXR but NO TST — Participants will receive symptom screening and CXR. No TST will be performed. If CXR abnormal or symptom positive, they undergo microbiological investigation. If the CXR is normal, and/or microbiological investigations negative - they receive LTBI treatment as per national guidelines. If microbiological investigation is positive they will be offered treatment for active TB.
  Arms: CXR for all/NoTST

SUMMARY:
The objective of the study is to compare outcomes from three different strategies for the management of household (HH) contacts of individuals with newly diagnosed microbiologically confirmed active pulmonary TB. The study is a cluster randomized trial with three arms of equal size. The first eligible member of the HH who provides signed informed consent to participate will be randomized to one of the three strategies. The three different study arms are as follows:

1. Standard care (control arm): Participants will receive symptom screening and tuberculin skin testing (TST). If symptom screen positive and/or TST positive, they undergo chest x-rays (CXR). If CXR abnormal, they undergo microbiological investigation. If CXR normal or if microbiological investigation negative, TST positive receive latent TB infection (LTBI) treatment. If microbiological investigation is positive, they will be offered treatment for active TB. For children under 5 years of age in Brazil, sputum induction will be performed for bacteriological investigation
2. GeneXpert (GX): Participants follow an algorithm similar to the standard care, however participants with positive symptom screen and/or positive TST will receive GX (i.e., GX replaces CXR in standard care algorithm). GX positive are considered to have active TB. TST positive and GX negative receive LTBI treatment. If an individual is not able to provide sputum, they will undergo a CXR.
3. CXR for all/NoTST: Participants will receive symptom screening and CXR. No TST will be performed. If CXR abnormal or symptom positive, they undergo microbiological investigation. If the CXR is normal, and/or microbiological investigations negative - they receive LTBI treatment as per national guidelines. If microbiological investigation is positive they will be offered treatment for active TB.

The study population includes HIV uninfected persons aged 5-50 years who are HH contacts of individuals with newly diagnosed microbiologically confirmed active pulmonary TB. The planned number of household contacts to recruit is about 1434 in total, or about 455 for each of the three arms. The study will take place in Benin and Brazil.

The primary study outcome is, of those eligible for LTBI therapy, the proportion starting therapy within 3 months of the index TB patient starting active TB treatment. Secondary outcomes measured in each study arm include societal costs, prevalence of microbiologically confirmed and clinically diagnosed active TB, prevalence of TB infection, Incidence of adverse events, proportion who complete LTBI therapy, sensitivity and specificity of Chest Xray reading in each study side, and prevalence of active TB diagnosed using CXR in participants who cannot produce a sputum sample. Details of the statistical analysis plan for each primary and secondary outcome are provided below. Applicable for Brazil only: To evaluate the applicability and performance of material for bacteriological investigation obtained from induced sputum in children under 5 years of age.

Study participants will be recruited over 18 months. Participants will be followed until LTBI treatment is completed.

DETAILED DESCRIPTION:
Background:

At a recent United Nations high level conference on TB a target was set that more than 30 million individuals should be treated for LTBI over the next 5 years. This ambitious goal will require massive scaling up of LTBI diagnosis and treatment - which will be challenging, if not impossible, with current approaches to diagnosis and treatment of latent TB. Two aspects of management of LTBI - need for CXR and need for TST - are controversial, as both can create important barriers to LTBI initiation, thereby reducing the individual as well as public health benefits of treatment. For TST, difficulties in training and quality assurance of administration and reading, and a global shortage of tuberculin material have reduced uptake. CXR was recommended by WHO in its 2018 guidelines for LTBI management as part of investigations to rule our active TB, however CXR services are not accessible in many settings and even if accessible, the cost for a CXR often falls on patients and is often prohibitively expensive. An alternate strategy is to use GeneXpert equipment, with the Xpert MTB/Rif test (hereafter labelled GX) to replace CXR to exclude prevalent active TB.

Study Objectives:

To compare outcomes from three different strategies for the management of HIV uninfected persons aged 5-50 years who are HH contacts of newly diagnosed microbiologically confirmed active pulmonary TB. (0-5 years only in Brazil)

Design:

This will be a cluster randomized trial with three arms of equal size; clusters will be defined as all the household contacts of patients with newly diagnosed active pulmonary TB. The first eligible member of the HH who provides signed informed consent to participate will be randomized to one of the three strategies. All subsequently enrolled members of the same HH will be assigned to the same study arm.

Study participants will be randomized to one of three different study arms:

1. Standard care (control arm): Participants will receive symptom screening and tuberculin skin testing (TST). If symptom screen positive and/or TST positive, they undergo chest x-rays (CXR). If CXR abnormal, they undergo microbiological investigation. If CXR normal or if microbiological investigation negative, TST positive receive latent TB infection (LTBI) treatment. If microbiological investigation is positive, they will be offered treatment for active TB. For children under 5 years of age in Brazil, sputum induction will be performed for bacteriological investigation.
2. GeneXpert (GX): Participants follow an algorithm similar to the standard care, however participants with positive symptom screen and/or positive TST will receive GX (i.e., GX replaces CXR in standard care algorithm). GX positive are considered to have active TB. TST positive and GX negative receive LTBI treatment. If an individual is not able to provide sputum, they will undergo a CXR.
3. CXR for all/NoTST: Participants will receive symptom screening and CXR. No TST will be performed. If CXR abnormal or symptom positive, they undergo microbiological investigation. If the CXR is normal, and/or microbiological investigations negative - they receive LTBI treatment as per national guidelines. If microbiological investigation is positive they will be offered treatment for active TB.

Population and Setting:

HIV uninfected persons aged 5-50 years who are household contacts newly diagnosed microbiologically confirmed active pulmonary TB can participate in the study. The planned number of household contacts to recruit is about 1434 in total, or about 455 for each of the three arms. The study will take place in five cities in two countries: Benin (Cotonou and Porto Novo) and Brazil (Rio de Janeiro, Manaus and Porto Alegre). In each city clinics will be selected that are representative of the diagnostic facilities and capacities available in most clinics in the country. For Brazil only they will include under 5 HIV uninfected.

Study duration:

Study participants will be recruited over a period of 18 months. Participants will be followed until LTBI treatment is completed (4-6 months depending on what treatment is given)

Outcomes:

Primary Outcome:

Of those eligible (measured or estimated) for LTBI therapy, the proportion starting therapy within 3 months of the index TB patient starting active TB treatment.

Secondary outcomes:

1. Societal costs (health system and patient costs) of the full cascade of care - from initial identification to LTBI therapy completion.
2. Prevalence of microbiologically confirmed and clinically diagnosed active TB - detected as part of the initial contact investigation, who initiate LTBI treatment within 3 months of the index TB patient starting active TB treatment.
3. Prevalence of positive TST (>5 mm or >10 mm) - overall, and by age group.
4. Incidence of grade 1-4 adverse events related to LTBI therapy.
5. Proportion who complete LTBI therapy - defined as having taken at least 80% of doses in 120% of allowed time.
6. Sensitivity and specificity of CXR reading by usual providers in each study site (reference standard will be readings by external reviewers).
7. Prevalence of active TB diagnosed using CXR in participants who cannot produce a sputum sample.
8. Applicable for Brazil only: To evaluate the applicability and performance of material for bacteriological investigation obtained from induced sputum in children under 5 years of age.

Statistical analyses:

Primary analysis The primary outcome is the proportion starting LTBI therapy of those eligible (measured or estimated) for latent TB therapy. 'Eligible' will be defined as: aged 5-50 years, HIV uninfected and TST >5mm. For the no TST arm, the expected prevalence for HIV uninfected HH contacts aged 5 years and older will be estimated from age-specific prevalence of positive TST among HH contacts tested in the other two arms. This expected prevalence will be used to estimate the proportion 'eligible' for LTBI therapy in the no TST arm. Treatment initiation will be defined as being given a prescription for LTBI therapy, or dispensed the first month of pills needed for LTBI therapy. Since this is a dichotomous outcome, the primary analysis will be a logistic regression, using an identity link, and estimated via generalized estimating equations (GEE) to account for clustering by household. An exchangeable correlation structure and empirical standard errors will be used. The proportion starting LTBI therapy within 3 months of the index TB patient starting active TB treatment will be compared in each experimental arm against the standard arm.

Secondary analyses.

1. Societal costs (health system and patient costs) of the full cascade of care - from initial identification to LTBI therapy completion will be considered. Using all relevant cost components and an ingredients approach, differences in health system costs will be assessed for each of the strategies. Patient time will be valuated based on an assumption of income equivalent to the average per capita income in the country. Health care personnel time will be valuated based on average salaries from information provided by facility management in each setting.
2. Prevalence of microbiologically confirmed and clinically diagnosed active TB - detected as part of the initial contact investigation, who initiate LTBI treatment within 3 months of the index TB patient starting active TB treatment, will be compared between all three arms.
3. Prevalence of positive TST (5 mm or 10 mm cut-points) by age group - 0-4 (for Brazil only), 5-10, 11-17, 18-24, 25-34 years, and older in Standard and GX Strategies. This is simple descriptive analysis - and will be presented as overall prevalence in the specified age groups, plus stratified by country.
4. Incidence of serious adverse events related to LTBI therapy. Adverse events are relatively rare dichotomous outcomes. As such, Poisson regression will be used to compare the occurrence of the adverse events between each of the two experimental arms and the conventional arm. To account for clustering by household, GEE, with an exchangeable correlation structure and empirical standard errors will be used. Investigators will compare in the same way - the occurrence of grade 1-2 adverse events reported by study investigators.
5. Completion of LTBI therapy - defined as taking at least 80% of doses in 120% of allowed time. (For 6H this means taking at least 144 doses within 216 days; for 4R this means 96 doses within 144 days, and for 3HR - 72 doses within 108 days.) Since this is a dichotomous outcome, the primary analysis will use logistic regression, with an identity link, and estimated via GEE to account for clustering by household. An exchangeable correlation structure and empirical standard errors will be used. The proportion completing treatment in each experimental arm against the standard arm will be compared.
6. Sensitivity and specificity of CXR reading by usual providers in each study site. For this analysis, the reference standard will be the readings by the external CXR review.
7. Active TB - defined as treatment initiated for active TB - detected only as a result of the CXR done in persons who could not produce a sputum sample.

ELIGIBILITY:
Inclusion Criteria:

* Index TB patients:

  1. New diagnosis of pulmonary microbiologically confirmed (smear, GX or culture) active TB within 30 days of treatment initiation.

     For Brazil: a new diagnosis of clinically pulmonary active is eligible.
  2. Must have at least one identified household contact, and HHC investigation has not been started already.
  3. Must agree to allow research team to access their medical history and approach their household contacts.
* Household contacts:

  1. Age 5-50 years for Benin and Age 0-50 for Brazil
  2. On average in the past 3 months - slept in the same house, at least one night per week, or spent at least one hour per day for 5 days per week.
  3. Pregnant woman can be included.
  4. People with prior active TB or latent TB therapy will be included. These participants will be assessed for prevalent active TB, although they will not be treated for LTBI. Hence they will be included in the analyses of yield of active case finding, but excluded from analyses of numbers diagnosed and treated for LTBI.

Exclusion Criteria:

* Index TB patients:

  1. Known drug-resistant TB (INH resistant, multidrug resistance or rifampin resistance) may be excluded - after discussion in each country with TB program officials. If the TB programme's policy is to screen contacts of MDR cases for active TB only and not provide any LTBI therapy, then index TB patients with MDR will be excluded as well as their HHCs. However, if the national TB program policy is to treat such individuals with standard LTBI therapy (since some HHCs of MDR patients will develop TB with drug-sensitive isolates later), then these index TB patients and their HHCs will be eligible. Hence, this will be a country-specific exclusion criterion.
  2. Index TB patient with previous history of active TB (because their HHC may have undergone investigation before - which may change their need for study interventions, and also potentially change their perceptions and behaviours in the study).
  3. Only has extra-pulmonary TB.
  4. No identified household contacts.
* Household contacts:

  1. Members of the household, but do not meet the minimum time definitions for HH contacts.
  2. Had TST/IGRA within 3 months.
  3. Had a CXR on the same day or after the date of diagnosis of the index TB patient.
  4. People living with HIV. (In most TB programs, HH contacts have unknown HIV status; HIV testing is recommended by WHO only if the index TB patient is known to have HIV co-infection). Contacts will be asked if they have been previously diagnosed to have HIV infection, and also asked if they are taking anti-retroviral therapy (if patients are receiving any medications, these will be checked carefully to verify what these are, and in particular if they are on anti-retroviral therapy). Both questions will be asked because some patients may be on therapy, but are not aware of the indication, or they may not wish to divulge their HIV status. If HHC are on anti-retroviral therapy and/or provide a history of previous HIV diagnosis, then they will be excluded, because the WHO recommended algorithm for investigation of household contacts who are HIV infected is different from that followed in the study arms. All index TB patients should undergo HIV testing based on national algorithm. If the index TB patient is found to be HIV positive, partner notification services will be recommended to the person living with HIV. The children of women who are HIV-infected should also undergo HIV testing. HIV testing will be offered to all household contacts who have not been HIV-tested within the last 6 months. If any household contact is found to be HIV-infected, they will be excluded pre-randomization. If there is a significant delay between identification of the household contacts and obtaining the HIV result, the HHCs can be randomized and then excluded post-randomization. These HHCs will be excluded from the modified intention to treat analysis, which will be the primary analysis. All HHCs identified to have HIV-infection will undergo investigations and treatment following WHO guidelines for HIV-infected household contacts.
  5. If one member family refuses to participate to the study and has no objection to have the other HH members to participate in the study, then we can proceed with the consent process with the other HHC. But if one household contact refuses to participate and objects to other HH members to take part of the study, then none of the HHC in this family can participate in the study. It is not necessary that all of the HHC signed consent but simply that no one objects. At any time a participant can refuse any test, or have other investigations - as ordered by their doctor/nurse or if they prefer).

Ages: 5 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1589 (Actual)
Dates: Start 2020-01-31 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
proportion starting therapy within 3 months of the index TB patient starting active TB treatment | LTBI treatment initiation within 3 months of the index TB patient starting active TB treatment.
  Of those eligible (measured or estimated) for LTBI therapy, the proportion starting therapy within 3 months of the index TB patient starting active TB treatment.

SECONDARY OUTCOMES:
Societal costs (health system and patient costs) of the full cascade of care | from the time of randomization until the end of investigations or the end of the second month of TB related treatment
  Societal costs (health system and patient costs) of the full cascade of care - from initial identification to LTBI therapy completion.
Prevalence of microbiologically confirmed and clinically diagnosed active TB | at baseline
  Prevalence of microbiologically confirmed and clinically diagnosed active TB - detected as part of the initial contact investigation, who initiate LTBI treatment within 3 months of the index TB patient starting active TB treatment.
Prevalence of positive TST (>5 mm or >10 mm) | at baseline
  Prevalence of positive TST (>5 mm or >10 mm) - overall, and by age group.
Incidence of grade 1-4 adverse events related to LTBI therapy. | from treatment initiation until the end of treatment case report form (CRF) has been completed
  Incidence of grade 1-4 adverse events related to LTBI therapy.
Proportion of participants who complete LTBI therapy | Approximately 4 to 6 months after treatment initiation (depending on regimen used)
  Completion of LTBI therapy - defined as having taken at least 80% of doses in 120% of allowed time.
Sensitivity and specificity of CXR | at baseline
  Sensitivity and specificity of CXR reading by usual providers in each study site (reference standard will be readings by external reviewers).
Prevalence of active TB diagnosed using CXR in participants who cannot produce a sputum sample. | at baseline
  Prevalence of active TB diagnosed using CXR in participants who cannot produce a sputum sample.
The outcome measure of performance is the percentage of patients with valid specimens obtained by the induction of sputum over all patients with indication for this technique. | at baseline
  Applicable for Brazil only: The outcome measure of performance is the percentage of patients with valid specimens obtained by the induction of sputum over all patients with indication for this technique.

CONTACTS AND LOCATIONS:
Overall Officials: Dick Menzies, Principal Investigator — RI-MUHC
Locations (4):
- Centre National Hospitalier Universitaire de Pneumo Phtisiologie de Cotonou (CNHU-PPC), Cotonou, Benin
- Brazil (3):
  - Manaus, Manaus
  - Porto Alegre, Porto Alegre
  - Centro de Estudos, Pesquisa e Desenvolvimento Tecnológico em Saúde Coletiva - CEPESC, Rio de Janeiro

REFERENCES:
- [Derived] Adjobimey M, Trajman A, Bastos ML, Valiquette C, Gibson D, Djohoun F, Oxlade O, Fregonese F, Affolabi D, Kouchade V, Aguiar E, Spener-Gomes R, Cordeiro-Santos M, Stein RT, Scotta M, Benedetti A, Menzies D. Rapid molecular testing or chest X-ray or tuberculin skin testing for household contact assessment of tuberculosis infection: A cluster-randomized trial. PLoS Med. 2025 Jul 28;22(7):e1004666. doi: 10.1371/journal.pmed.1004666. eCollection 2025 Jul. PMID 40720526
- [Derived] Trajman A, Adjobimey M, Bastos ML, Valiquette C, Oxlade O, Fregonese F, Affolabi D, Cordeiro-Santos M, Stein RT, Benedetti A, Menzies D. GeneXpert or chest-X-ray or tuberculin skin testing for household contact assessment (GXT): protocol for a cluster-randomized trial. Trials. 2022 Aug 2;23(1):624. doi: 10.1186/s13063-022-06587-0. PMID 35918722

DOCUMENTS (2):
  • Study Protocol (2022-03-14): https://cdn.clinicaltrials.gov/large-docs/23/NCT04528823/Prot_002.pdf
  • Informed Consent Form (2019-06-03): https://cdn.clinicaltrials.gov/large-docs/23/NCT04528823/ICF_000.pdf